CLINICAL TRIAL: NCT05312541
Title: A Comparative Study Between Analgesic Effect of Opioid Free and Opioid Based General Anesthesia Technique in Patients Undergoing Open Radical Nephrectomy Surgery.A Prospective Randomized Controlled Trial
Brief Title: A Comparative Study Between Analgesic Effect of Opioid Free and Opioid Based Anesthesia in Radical Nephrectomy Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed nabih youssef, Lecturer of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-2-2022
Record Dates: First submitted 2022-03-12; First posted 2022-04-05 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Opioid Free Anesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomization will be done by computer generated numbers and concealed by serially numbered, opaque and sealed envelopes. The details of the series will be unknown to the investigators and the group assignment will be kept in asset of sealed envelopes each bearing only the case number on the outside. Prior to surgery the appropriate numbered envelopes will be opened by the nurse, the card inside will determine the patient group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid Based Anesthesia (Placebo Comparator): Pre induction of general anesthesia with placebo 1 h before surgery. induction of general anesthesia with fentanyl1ug/kg/ iv then infusion of 1 ug/kg/h
  Interventions: Procedure: pre emptive local anaesthetic wound infiltration
- opioid free anesthesia (Active Comparator): Pre induction of general anesthesia with gabapentin 300 mg tab 1 h before surgery. induction of general anesthesia with ketamine 0.5 mg/kg iv, Lidocaine 1 mg/kg iv then continuous infusion with 2 mg/kg/hr, dexamethasone 0.1 mg/kg.iv, magnesium sulfate 20 mg/kg.iv
  Interventions: Procedure: pre emptive local anaesthetic wound infiltration

INTERVENTIONS:
Procedure: pre emptive local anaesthetic wound infiltration — Before skin incision by 15 min the surgeon will infiltrate the wound by syringe containing 20 ml mixture of (10 ml xylocaine 2%and 10 ml bupivacaine 0. 5%) in both groups
  Other Names: xylocaine and bupivacaine local anaesthetic mixture

SUMMARY:
Patients undergoing nephrectomy have a high incidence of postoperative pain. In the perioperative period, these patients are often treated with patient-controlled opioids, epidural analgesia, or both. While effective, both of these treatment modalities carry risk, ie, opioids have a side effect profile including pruritus, nausea,vomiting, increase the risk of oversedation and apnea in patients at risk (eg, those with sleep apnea), difficulty in voiding, and ileus. These complications may lead to a prolonged hospital stay. High dose opioids can also cause acute opioid tolerance and hyperalgesia. Epidurals have been associated with hypotension, post dural puncture headaches, changes in management of anticoagulation Opioid free anesthesia (OFA) is a technique in which no intraoperative opioid administered through any route, including systemic, neuraxial, or tissue infiltration.Opioid free anesthesia has many advantages especially avoiding opioid overdose and opioid-induced hyperalgesia. The most important advantage of OFA seems to be the potential improvement of recovery profile in obese patients. OFA depends on combinations of non-opioid agents and adjuncts, including propofol, lidocaine, magnesium, dexmedetomidine, and ketamine to produce anesthesia, and analgesia.

Aim of the work our study aim to compare the analgesic effect of OFA and opioid based general anesthesia using pre emptive wound infiltration in patients undergoing open radical nephrectomy surgery.

Objectives:

1. To evaluate analgesic effect of each group intra operative {heart rate, and systolic and diastolic blood pressure }
2. To evaluate analgesic effect of each group post operative [total opioid consumption in 24h postoperative , Postoperative VAS , hemodynamic).
3. To estimate the incidence of early postoperative complication in both groups

DETAILED DESCRIPTION:
This a randomized control trial is designed to include (74) patients ASA physical status II patients ranging from(18) to(70)years old scheduled for open radical nephrectomy

Patients meeting the inclusion criteria will be randomly assigned to receive either :

Group I :Opioid Based Anesthesia (n=37) GroupII: Opioid Free Anesthesia:(n=37) Anesthesia management

Preoperative procedures:

Full history and investigation will be taken in the form of complete blood count , blood sugar,liver function tests. Kidney function tests ,electrolytes and coagulation profile. Pre induction of general anesthesia with gabapentin 300 mg tab or placebo 1 h before surgery while gabapentin in (Opioid free Anesthesia) and placebo in (Opioid Based Anesthesia) . After securing IV access by 20G cannula, all patients will receive 0.05mg/kg midazolam for anxiety. Ranitidine 50mg, metoclopramide 10mg and antibiotic 50mg/kg as a premedication.Intraoperative monitoring includes ASA standard monitoring Electrocardiography (ECG), noninvasive blood pressure, pulse oximetry for O2 saturation, end-tidal carbon dioxide (CO2) values by capnography.

Intraoperative procedures:

Induction of general anesthesia in both groups will be done by 2mg \kg propofol, and 0.5mg\kg atracurium. to facilitate endotracheal intubation, with fentanyl1ug/kg/ iv then infusion of 1 ug/kg/h in group I (Opioid Based Anesthesia) and with ketamine 0.5 mg/kg iv, Lidocaine 1 mg/kg iv then continuous infusion with 2 mg/kg/hr, dexamethasone 0.1 mg/kg.iv, magnesium sulfate 20 mg/kg.iv in group II (Opioid Free Anesthesia) after induction.

Anesthesia maintenance will be achieved in both group with endotracheal tube (ETT) with suitable size, 1.2 minimium alveolar concentration of isoflurane, volume controlled mode ventilation, respiratory rate will be adjusted according to Et CO2 to range between 35-40 mmHg, a tidal volume of 6-8 ml/kg and mixture of gases in proportion 50% oxygen and 50% air, with positive end expiratory pressure (PEEP) 5 cm H2O and0.1 mg\kg atracurium every 30 min.

Intervention Before skin incision by 15 min the surgeon will infiltrate the wound by syringe containing 20 ml mixture of (10 ml xylocaine 2%and 10 ml bupivacaine 0. 5%) in both groups. By the end of surgery, anaesthesia will be discontinued ,patient will be reversed by neostigmine 0.05mg\kg and atropine0.02mg\kg, extubation will be done and patient will be transferred to post anaesthesia care unit (PACU).

Postoperative

1. The pain assessment after full recovery will be performed using a 10 cm visual analog scale (VAS) (0- no pain and 10 cm maximum pain) .Postoperative pain assessments using VAS at 0 point (the full recovery state which is defined as a state of consciousness of individual when he is awake or easily arousable and aware of his surroundings and identity, 2 hr, 6 hr, 12 hr, and at 24 hr. IV paracetamol 1 g every 6 hours will be administered for both groups.

   The time to first request of postoperative analgesic is defined as( the time interval from tracheal extubation to first dose of morphine adminstration) will be recorded .Rescue postoperative analgesic will be administrated if VAS ≥ 4 at rest or on patient's demand with IV morphine sulphate 0.03 mg/kg with maximum dose 20 mg per day in both groups .the total amount of morphine in the first postoperative 24 hours will be calculated in both groups.
2. Post operative hemodynamic will be assessed(heart rate ,systolic and diastolic blood pressure at the same time point)
3. Incidence of complication will be assessed:

   * Nausea and vomiting
   * Respiratory complications(bronchospasm , laryngospasm , respiratory depression)

Measurement tools

1. Patients demographic data will be collected; age, gender, and duration of anesthesia
2. Intraoperative hemdynamic (Heart rate ,systolic and diastolic blood pressure).
3. Postoperative pain assessments using VAS at at 0 point (the full recovery state), 2 hr, 6 hr, 12 hr, and at 24 hr
4. Time to first request of rescue postoperative analgesic
5. Total opioid consumption in 24 h postoperative
6. Postoperative hemdynamic (Heart rate ,systolic and diastolic blood pressure at the same time point)

ELIGIBILITY:
Inclusion Criteria:

1. Gender both males and females
2. ASA Class II
3. Age 18-70 years
4. Patients undergoing open radical nephrectomy

Exclusion Criteria:

1. Allergy to local anesthetic
2. Infection of the skin at the site of local infiltration
3. Cvs problem(ischemic heart disease,arrhythmias{heart block, supraventricular tachyarrhythmia (SVT),atrial fibrillation (AF),multiple extra systole)
4. Liver and renal impairment(elevated liver enzymes (ALT, AST two to three fold), chronic renal failure (CRF) )

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
The Time to first request of opioid analgesia | it will be measured from tracheal extubation to first request of postoperative analgesia in the first 24 hours postoperative and it will be expressed in minutes
  the time interval between tracheal extubation and the first request to postoperative analgesia

SECONDARY OUTCOMES:
Total opioid consumption | the total amount of morphine in the first postoperative 24 hours will be calculated
  total amount of morphine in the first postoperative 24 hours
Postoperative VAS score | Postoperative pain assessments using VAS at 0 point (the full recovery state ), 2 hours, 6 hours, 12 hours,and at 24 hours postoperative.
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

CONTACTS AND LOCATIONS:
Overall Officials: Heba ismail, professor, Study Director — Anesthesia department , Cairo university
Locations (1):
- Kasr Alainy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No